CLINICAL TRIAL: NCT06717126
Title: A Phase II, Multi-centre, Open Label, Randomised Study to Evaluate the Anti-tumour Activity of Roginolisib in Patients With Advanced/Metastatic Ocular/Uveal Melanoma
Brief Title: A Randomised Phase II Study of Roginolisib in Patients With Advanced/Metastatic Uveal Melanoma
Acronym: OCULE-01
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: iOnctura (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOA-244-201
Record Dates: First submitted 2024-11-18; First posted 2024-12-04 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Uveal Melanoma; Ocular Melanoma
Keywords: Uveal; Ocular; Melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma

STUDY DESIGN:
Intervention Model Description: Randomised parallel-arm, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 - Roginolisib 80mg (Experimental): IOA-244: 80 mg (corresponding to 72 mg roginolisib) daily
  Interventions: Drug: roginolisib
- Arm 2 - Investigator choice of standard of care (Active Comparator): Investigator´s choice of therapy
  Interventions: Drug: Investigator choice of standard therapy
- Arm 3 - Roginolisib 40mg (Experimental): IOA-244: 40 mg (corresponding to 36 mg roginolisib) daily
  Interventions: Drug: roginolisib

INTERVENTIONS:
Drug: roginolisib — rognolisib
  Other Names: IOA-244
  Arms: Arm 1 - Roginolisib 80mg; Arm 3 - Roginolisib 40mg
Drug: Investigator choice of standard therapy — Investigator will choose the most appropriate treatment standardly given to patients
  Arms: Arm 2 - Investigator choice of standard of care

SUMMARY:
The goal of this clinical trial is to learn how roginolisib works in comparison to standard treatment in adult patients with uveal/ocular melanoma. The main questions it aims to answer are:

Does roginolisib extend overall survival compared to standard treatment? How does dosing of roginolisib impact quality of life compared to standard treatment?

DETAILED DESCRIPTION:
A Phase II open-label, randomised, parallel-arm study, which will assess the clinical efficacy of oral roginolisib (IOA 244 [roginolisib hemi-fumarate]) as monotherapy against a control of Investigator´s treatment choice in patients with advanced or metastatic uveal melanoma (UM).

This study will enrol approximately 85 male and female patients aged over 18 years with advanced or metastatic UM, who have progressed following at least 1 prior immunotherapy treatment. The disease must be measurable (i.e., at least 1 measurable lesion) as per RECIST v1.1 by Computerised Tomography (CT) scan or Magnetic Resonance Imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or older;
2. Histologically or cytologically proven diagnosis of advanced or metastatic UM or ocular melanoma (arising from ocular melanocytes regardless of intraocular location)
3. Patients who have progressed following at least 1 prior immunotherapy treatment for advanced or metastatic UM. For patients who are HLA-A*02:01 positive prior treatment should have included tebentafusp, if available or patients clinically suitable. Patients who have also received prior melphalan hepatic infusion may be included;
4. Presence of at least one lesion suitable for biopsy. Biopsies will be mandatory at Screening and C5D1 (see Sections 8.1.3 and 8.6 for more information);
5. Presence of at least one measurable lesion as per RECIST v1.1. Any lesion that is biopsied cannot be used as a measurable lesion for the purposes of RECIST v1.1 assessments;
6. ECOG performance status of 0 to 1;
7. Male or female patients of child-bearing potential must be willing to use highly effective forms of contraception (refer to APPENDIX 7 for details on highly effective methods of contraception and definitions of women of childbearing potential and of fertile men)
8. All other relevant medical conditions must be well managed and stable, in the Investigator's opinion, for at least 28 days prior to first dose of roginolisib;
9. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.

Exclusion Criteria:

1. Inability to swallow oral medication;
2. a). History of a prior Grade 3 or 4 irAE or any grade ocular irAE from prior immunotherapy which did not respond to corticosteroid therapy or resolved with treatment interruptions and returned to at least Grade 1; b). Have not recovered from toxic effect(s) of prior therapy to ≤ Grade 1, other than alopecia or fatigue or neuropathy which must be ≤ Grade 1;
3. Presence of symptomatic or untreated CNS metastases or CNS metastases that require doses of corticosteroids within the prior 3 weeks to first dose of roginolisib. Patients with brain metastases are eligible if lesions have been treated with localised therapy and there is no evidence of progressive disease for at least 4 weeks prior to the first dose of IMP;
4. Abnormal liver enzymes defined as:

   1. ALT or AST ≥ 3× upper limit of normal (ULN) (≥ 5× ULN in patients with liver metastases);
   2. Total bilirubin ≥ 1.5 × ULN are excluded unless direct bilirubin is ≤ ULN. If there is no institutional ULN, then direct bilirubin must be < 40% of total bilirubin to be eligible (except patients with Gilbert syndrome);
5. Any other clinically significant out of range laboratory values;
6. Clinically significant cardiac disease or impaired cardiac function which may limit the patient´s participation in the clinical study. These may include unstable angina (i.e., not responsive to medical intervention), myocardial infarct in last 6 months, QTcF prolongation of more than 500 ms;
7. Evidence of interstitial lung disease or active, non-infectious pneumonitis, pulmonary fibrosis;
8. Active infection requiring systemic antibiotic therapy. Patients requiring systemic antibiotics for infection must have completed therapy at least 1 week prior to the first dose of IMP;
9. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection per institutional protocol;
10. Malignant disease, other than that being treated in this study (e.g., skin/cutaneous and/or mucosal melanoma). Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to first dose of IMP; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type;
11. Any medical condition that would, in the Investigator's or Sponsor's judgment, prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results;
12. Treatment with anti-tumour medications or investigational drugs within 14 days or 5 half-lives (whichever is longer) of administration of first dose of IMP;
13. Major surgery within 2 weeks of the first dose of IMP (minimally invasive procedures such as bronchoscopy, tumour biopsy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery and are not exclusionary);
14. Radiotherapy within 4 weeks of the first dose of IMP, with the exception of palliative radiotherapy to a limited field, such as for the treatment of bone pain or a focally painful tumour mass;
15. Pregnant, likely to become pregnant, or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Patients will be followed up for overall survival every 12 weeks, for 96 weeks from last patient enrolled, until their death or end of the study
  To evaluate clinical efficacy of roginolisib as single agent, against Investigator's choice of therapy by assessment of overall survival (OS)

SECONDARY OUTCOMES:
Progression free survival (PFS) | Patients will be followed up for progression free survival every 8 weeks, for 96 weeks from last patient enrolled, until progression of disease, their death or end of the study
  PFS measured from the time from the date of the first dose of IMP until the earliest date of disease progression as determined by radiographic/objective disease assessment as per RECIST v1.1
Objective response rate (ORR) | Every 8 weeks whilst on treatment anticipated to be 52 weeks
  ORR defined as percentage of patients with a Complete Response (CR) or Partial Response (PR)
Duration of response (DOR) | Every 8 weeks up to 96 weeks from start of treatment
  DOR defined as the time from the date of first documented response (CR, PR) by RECIST v1.1 until the date of documented progression or death in the absence of disease progression
Time to response | Every 8 weeks whilst on treatment anticipated to be 52 weeks
  Time to Response is defined as the time from date of first dose of IMP until the date of first documented objective response
Disease control rate (DCR) | Every 8 weeks whilst on treatment anticipated to be 52 weeks
  DCR is defined as the proportion of patients with a Best Objective Response (BOR) of CR or PR or Stable disease (SD) recorded at ≥8 weeks (±1 week),
Clinical benefit rate (CBR) | Measured at Cycle 5 - approximately 16 weeks from start of dosing
  CBR is defined as the proportion of patients with a BOR of CR or PR or SD recorded at Cycle 5 Day 1
Safety and tolerability | Every 4 weeks whilst on treatment anticipated to be 52 weeks
  Assessed by AEs, laboratory parameters, vital signs, physical exam, ECG and ECOG status
Pharmacokinetics (PK) | Every 4 weeks for 52 weeks from start of treatment
  Concentration of roginolisib at pre-dose and steady state levels (including Area under the curve [AUC], population PK)
Safety of 40 vs 80 mg of roginolisib | Every 4 weeks whilst on treatment anticipated to be 52 weeks
  Assessed by AEs, laboratory parameters, vital signs, physical exam, ECG and ECOG status
Health care utilisation | Every 4 weeks whilst on treatment anticipated to be 52 weeks
  Assessed by health resource used
Quality of Life | Every 4 weeks for 52 weeks from start of treatment
  Changes in Patient Reported Outcomes (PRO) relative to baseline. Patients to complete EuroQoL Research Foundation EQ-5D-5L Health questionnaire
Quality of Life | Every 4 weeks for 52 weeks from start of treatment
  Changes in Patient Reported Outcomes (PRO) relative to baseline. Patients to complete European Organisation for Research and Treatment of Cancer (EORTC QlQ-C30)
Quality of Life | Every 4 weeks for 52 weeks from start of treatment
  Changes in Patient Reported Outcomes (PRO) relative to baseline. Patients to complete Epworth Sleepiness Scale (ESS) questionnaire
Quality of Life | Every 4 weeks for 52 weeks from start of treatment
  Changes in Patient Reported Outcomes (PRO) relative to baseline. Patients to complete Fatigue Severity Scale (FSS)

OTHER OUTCOMES:
Circulating Tumour Deoxyribonucleic Acid (ctDNA) | Every 4 weeks for 52 weeks from start of treatment
  To assess any treatment-related changes in the pre and on treatment levels of circulating DNA from blood

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lahn, MD, Study Director — iOnctura
Locations (16):
- Italy (5):
  - SSD Tumori Rari e Melanoma Viale Orazio Flacco, Bari
  - IRCSS National Cancer Institute, "G.Pascale" Foundation Dip. CORP-S di Ricerca ed Assistenziale Cute, Melanoma lmmunologia Oncologica Sperimentale e Terapie Innovative, Napoli
  - IRCSS Istituto Oncologico Veneto UOS Oncologia 2 del Melanoma Ospedale Busonera, Padua
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - A.O.U.S. Santa Maria delle Scotte, Siena
- Spain (5):
  - Institut Catala d'Oncologia - ICO L'Hospitalet, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario Universitario de Santiago - CHUS, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, University of Seville, Seville
  - Consorcio Hospital General Universitario de València - CHGUV, Valencia
- United Kingdom (6):
  - East and North Hertfordshire NHS Trust (Mount Vernon Cancer Centre), Northwood, Middlesex
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral
  - Beatson West of Scotland Cancer Centre, Glasgow (NHS Greater Glasgow & Clyde), Glasgow
  - University College London Hospital NHS, London
  - Royal Marsden Hospital, London
  - University Hospital Southampton NHS Foundation, Southampton

IPD SHARING:
Plan to Share IPD: Undecided